CLINICAL TRIAL: NCT00551252
Title: A Phase II Study of the Association of Glivec® (Imatinib Mesylate, Formerly Known as STI 571) Plus Gemzar® (Gemcitabine) in Patients With Unresectable, Refractory, Malignant Mesothelioma Expressing Either PDGFR-Beta or C-Kit
Brief Title: A Phase II Study of the Association of Glivec® Plus Gemzar® in Patients With Unresectable, Refractory, Malignant Mesothelioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gruppo Italiano MEsotelioma (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMe/01/06
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2007-10-30 (Estimated); Status verified 2007-10

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Imatinib Mesylate; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental)
  Interventions: Drug: Imatinib mesylate plus Gemcitabine

INTERVENTIONS:
Drug: Imatinib mesylate plus Gemcitabine — Imatinib (400 mg daily) + Gemcitabine (500 mg/sqm, days 1 and 8 every 21 days) for a maximum of 6 cycles

SUMMARY:
The purpose of this study is to evaluate the antitumor activity of a combination of Imatinib mesylate and Gemcitabine in patients with unresectable malignant mesothelioma expressing either PDGFR-beta or C-kit

DETAILED DESCRIPTION:
TITLE "A phase II study of the association of Glivec® (Imatinib mesylate, formerly known as STI 571) plus Gemzar® (Gemcitabine) in patients with unresectable, refractory, malignant mesothelioma expressing either PDGFR-beta or C-Kit"

PURPOSE Primary objective of the phase II

> Efficacy, i.e., response rate to study drugs

Secondary objectives of the phase II

* Duration of response
* Time to progression
* Toxicity profile
* Overall survival

PRIMARY VARIABLE The primary efficacy variable for the phase II part of the study is Best Overall Tumor Response, evaluated using the "Modified RECIST criteria for assessment of response in malignant pleural mesothelioma"

SECONDARY VARIABLES

* Progression-free survival (PFS) form 1st administration onwards
* Overall survival
* Safety criteria, according to NCI-CTC criteria version 3.0

EFFICACY Objective tumor response assesed using the "Modified RECIST criteria for assessment of response in malignant pleural mesothelioma" SAFETY

* Adverse events
* Vital signs
* Clinical and biohumoral findings

TREATMENT SCHEDULE

* Gemzar 500 mg/m2, i.v., days 1 and 8 of a 21-days schedule, plus
* Glivec 400 mg/die., per os

STATISTICAL DESIGN The study follows a two-stage design, according to the Simon model. We assume that with a response rate of 5% (H0) or less the drug is likely to be ineffective, and also, that, for the drug to be effective, a target response rate of 15% (H1) is required. With a probability errors alfa of 5% and beta 20%, the calculated sample size is as reported in "PLANNED NUMBER OF PTS."

PLANNED NUMBER OF PTS. 23 or 56 patients, evaluable for efficacy. The number depends on the response rate. When 2 or more objective responses, i.e., CR or PR, are observed in the first 23 patients, the total number of patients will be increased to 56, otherwise the study will be stopped

STATISTICAL EVALUATION Efficacy and safety variables will be evaluated descriptively. Indeed, ORR estimates and its exact 95% confidence interval will be calculated. Kaplan-Meier method will be used to estimate duration of response, PFS and OS

DURATION OF TREATMENT All patients are scheduled to receive at least two cycles of chemotherapy unless there is unacceptable toxicity, progressive disease, or the patient requires or asks for withdrawal from the study Responding patients will receive treatment for 6 cycles or earlier if progression or unbearable toxicity Disease status will be re-evaluated every two cycles, using the same imaging procedures used at baseline, i.e., CT or NMR

INCLUSION CRITERIA

* Age of > 18 years and < 72 years
* Patients with a histologically proven malignant mesothelioma of the pleura or of the peritoneum, expressing either PDFGR-beta or C-Kit by immunochemistry (ICH)
* Locally advanced disease, unsuitable for curative surgical resection, or metastatic disease
* Confirmed progression of the disease according to modified REcist-criteria, documented after a first-line, systemic (premetrex+cisplatin regimen) or local treatment (i.e., intrapleuric)
* ECOG Performance Status of 0, 1 or 2
* Life expectancy of at least 3 months
* Capability of understanding the objectives of the study and giving written informed consent
* Willingness and ability to comply with study requirements
* Sufficient caloric and fluid intake, including patients under enteral or parenteral nutrition

EXCLUSION CRITERIA

* Co-existing tumors of different histologic origin, except non melanomatous localized skin cancer and/or in situ cervical carcinoma
* A history of earlier tumors of different histologic origin being in complete remission since less than 5 years
* Unresolved toxicity from prior antitumor treatment(s)
* Primary peritoneal mesothelioma
* Any of the following abnormal baseline hematological values:

  * Hb < 9 g/dL
  * WBC < 3 x 109/L
  * Neutrophils < 1.5 x 109/L
  * Platelets < 100 x 109/L
  * Serum bilirubin > 2.5 mg/dL
  * ALAT and ASAT > 3 x UNL (unless due to liver metastases)
  * Serum creatinine > 1.5 mg/dL
* Clinically relevant cardiovascular disease, i.e., myocardial infarction or other severe coronary artery diseases within the prior 6 months, cardiac arrythmia requiring medication, uncontrolled hypertension, overt cardiac failure or non compensated chronic heart disease in NYHA class II or more
* History of psychiatric disabilities, potentially interfering with the capability of giving adequate informed consent
* Pregnant or lactating women or inability/unwillingness to practice a medically approved method of contraception during study period (including 3 months following the end of treatment)
* Uncontrolled active infections
* Any condition which, in the judgement of the Investigator, would place the patient at undue risk or interfere with the results of the study

ELIGIBILITY:
Inclusion Criteria:

* Age of > 18 years and < 72 years
* Patients with a histologically proven malignant mesothelioma of the pleura or of the peritoneum, expressing either PDFGR-beta or C-Kit by immunochemistry (ICH)
* Locally advanced disease, unsuitable for curative surgical resection, or metastatic disease
* Confirmed progression of the disease according to modified REcist-criteria, documented after a first-line, systemic (premetrex+cisplatin regimen) or local treatment (i.e., intrapleuric)
* ECOG Performance Status of 0, 1 or 2
* Life expectancy of at least 3 months
* Capability of understanding the objectives of the study and giving written informed consent
* Willingness and ability to comply with study requirements
* Sufficient caloric and fluid intake, including patients under enteral or parenteral nutrition

Exclusion Criteria:

* Co-existing tumors of different histologic origin, except non melanomatous localized skin cancer and/or in situ cervical carcinoma
* A history of earlier tumors of different histologic origin being in complete remission since less than 5 years
* Unresolved toxicity from prior antitumor treatment(s)
* Primary peritoneal mesothelioma
* Any of the following abnormal baseline hematological values:

  * Hb < 9 g/dL
  * WBC < 3 x 109/L
  * Neutrophils < 1.5 x 109/L
  * Platelets < 100 x 109/L
  * Serum bilirubin > 2.5 mg/dL
  * ALAT and ASAT > 3 x UNL (unless due to liver metastases)
  * Serum creatinine > 1.5 mg/dL
* Clinically relevant cardiovascular disease, i.e., myocardial infarction or other severe coronary artery diseases within the prior 6 months, cardiac arrythmia requiring medication, uncontrolled hypertension, overt cardiac failure or non compensated chronic heart disease in NYHA class II or more
* History of psychiatric disabilities, potentially interfering with the capability of giving adequate informed consent
* Pregnant or lactating women or inability/unwillingness to practice a medically approved method of contraception during study period (including 3 months following the end of treatment)
* Uncontrolled active infections
* Any condition which, in the judgement of the Investigator, would place the patient at undue risk or interfere with the results of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2008-01; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Every two months

SECONDARY OUTCOMES:
Progression-free-survival; Overall Survival; Safety | Follow-up after end of treatment will be every three months; safety will be analyzed throughout the whole study

CONTACTS AND LOCATIONS:
Overall Officials: Camillo Porta, MD, Principal Investigator — Medical Oncology, IRCCS San Matteo University Hospital Foundation, pavia, Italy
Locations (1):
- Medical Oncology, IRCCS San Matteo University Hospital Foundation, Pavia, Italy

REFERENCES:
- [Background] Bertino P, Porta C, Barbone D, Germano S, Busacca S, Pinato S, Tassi G, Favoni R, Gaudino G, Mutti L. Preliminary data suggestive of a novel translational approach to mesothelioma treatment: imatinib mesylate with gemcitabine or pemetrexed. Thorax. 2007 Aug;62(8):690-5. doi: 10.1136/thx.2006.069872. Epub 2007 Feb 20. PMID 17311837
- See also: Italian Mesothelioma Group Homepage — http://www.gime.it